CLINICAL TRIAL: NCT05707728
Title: Evaluation of Role of Intraoperative Ultrasound in Gross Total Resection of Gliomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fadwa Ahmwd Ahmed, resident, Assiut University
Other Study IDs: intraoperative ultrasound
Record Dates: First submitted 2023-01-21; First posted 2023-02-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- totally resection of glioma using intraoperative ultrasound: totally resection of glioma using intraoperative ultrasound
  Interventions: Device: intraoperative ultrasound

INTERVENTIONS:
Device: intraoperative ultrasound — intraoperative cranial ultrasound

SUMMARY:
The use of intraoperative ultrasound (IOUS )seems to have significantly increased the Gross total Resection rate achieved in brain gliomas surgery. As regard intraoperative visualisation of the tumor and its residuals, the effectiveness of IOUS has been documented in a series of 192 High Grade glioma patients, in which the combination of neuronavigation and IOUS was also related to increased overall survival in a prospective study of 32 patients, documented a good level of agreement between intraoperative ultrasonography and postoperative contrast-enhanced MRI in detecting tumor residuel they concluded that the IOUS produces results similar to those of MRI, and therefore, can be used to maximize tumor resection.

DETAILED DESCRIPTION:
The use of intraoperative ultrasound (IOUS) during neurosurgical procedures was first described in 1978 by MH Reid The initial interest towards US as an imaging tool in neurosurgery progressively weaned from the 80's until the early 2000's in favor of other imaging techniques such as CT and MRI

Maximal safe resection represents the gold standard for surgery of malignant brain tumors:

gross total resection of the tumor while preserving the surrounding functional brain tissue is the main goal, since it is associated with longer survival and better patient quality of life This is particularly true for gliomas, the most common primary malignant brain tumors Concerning gross total resection, accurate localization and precise delineation of the tumor margins are required in order to avoid devastating lesions on nervous structures Ultrasound may provide an alternative tool to intraoperative magnetic resonance imaging (MRI) for delineating tumor Tissues and improving the chances of gross total resection The purpose of brain tumor removal is maximal resection while sparing healthy tissues. The extent of resection is a key prognostic factor in survival time, functional recovery, and tumor recurrence rates The optimal results of brain lesion surgery may be achieved by maximal surgical resection without disturbance of neurological functions Due to the imprecise correlation between preoperative images,intraoperative anatomy, and also poor differentiation of some tumors from a normal tissue, better delineation of normal from tumor tissue intraoperatively could improve clinical outcome as increasing chance of total resection and decreasing normal tissue damage . Intraoperative imaging technology increases the extent of tumor resection and patients' outcome including survival time.

Intraoperative MRI are time-consuming and of high cost. Computed tomography (CT) usually is not of choice as ionizing radiation and limited mass delineation. Several researches have demonstrated that the image quality of ultrasound has improved enough to visualize and guide tumor resection The most important disadvantage of neuronavigation is the inconsistency with preoperative images from changes of the lesion and critical anatomic structures associated with brain shift as intraoperative tumor resection or cerebrospinal fluid drainage. This creates the need for updating the preoperative image with the intraoperative image

The use of intraoperative ultrasound (IOUS )seems to have significantly increased the Gross total Resection rate achieved in brain gliomas surgery. As regard intraoperative visualisation of the tumor and its residuals, the effectiveness of IOUS has been documented in a series of 192 High Grade glioma patients, in which the combination of neuronavigation and IOUS was also related to increased overall survival in a prospective study of 32 patients, documented a good level of agreement between intraoperative ultrasonography and postoperative contrast-enhanced MRI in detecting tumor residuel they concluded that the IOUS produces results similar to those of MRI, and therefore, can be used to maximize tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with all grades of gliomas confirmed by MRI , MRI with contrast and MR spectroscopy .
* Age of the patient: any age.
* Both sex

Exclusion Criteria:

* • Other tumours and space occupying lesion (sol) rather than gliomas confirmed by histopathology and preoperative imaging

  * Patients unfit for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with all grades of gliomas confirmed by MRI any age and any sex
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients who have gliomas and totally resection by using intraoperative ultrasound | 1 year
  Numbers of patients who have gliomas and totally resection by using intraoperative ultrasound

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Giammalva, G.R.; Iacopino, D.G.; Azzarello, G.; Gaggiotti, C.; Graziano, F.; Gulì, C.; Pino, M.; Maugeri, R. End-of-Life Care in High-Grade Glioma Patients. The Palliative and Supportive Perspective. Brain Sci. 2018, 8, 125. [CrossRef] [PubMed] 2. La Torre, D.; Maugeri, R.; Angileri, F.F.; Pezzino, G.; Conti, A.; Cardali, S.M.; Calisto, A.; Sciarrone, G.; Misefari, A.; Germanò, A.; et al. Human leukocyte antigen frequency in human high-grade gliomas: A case-control study in Sicily. Neurosurgery 2009, 64, 1082-1088. [CrossRef] [PubMed] 3. Maugeri, R.; Schiera, G.; Di Liegro, C.M.; Fricano, A.; Iacopino, D.G.; Di Liegro, I. Aquaporins and brain tumors. Int. J. Mol. Sci. 2016, 17, 1029. [CrossRef] [PubMed] 4. Grasso, G.; Meli, F.; Fodale, V.; Calapai, G.; Buemi, M.; Iacopino, D.G. Neuroprotective potential of erythropoietin and darbepoetin alfa in an experimental model of sciatic nerve injury. J. Neurosurg. Spine 2007, 7, 645-651. [CrossRef] [PubMed] 5. Unsgaard G, Ommendal S, Muller T, Gronningsaeter A, Hernes TAN. Neuronavigation by intraoperative three-dimensional ultrasound: initial experience during brain tumor resection. Neurosurgery. 2002;50(4): 804-12. 6. Almenawer SA, Badhiwala JH, Alhazzani W, Greenspoon J, Farrokhyar F, Yarascavitch B, et al. Biopsy versus partial versus gross total resection in older patients with high-grade glioma: a systematic review and metaanalysis. Neuro Oncol. 2015;17(6):868-81. 7. Elserry TH, Anwer H, Radwan HA. Introduction of vaginal probe for intraoperative ultrasound of intra-axial brain lesions. Egyp J Neurosurg. 2013; 28(4):5-12. 8. Zhang ZZ, Shield LBE, Sun DA, Zhang YP, Hunt MA, Christopher BS. The art of intraoperative glioma identification. Front Oncol. 2015;5(175):1-7. 9. Gronningsaeter A, Kleven A, Ommedal S, Aarseth TE, Lie T, Lindseth F, Lango T, Unsgaar